CLINICAL TRIAL: NCT05195762
Title: 12-Week Clinical Study to Determine the Safety, Tolerability, and Clinical Effect of NFX-179 Gel in Subjects With Epidermal Nevi
Brief Title: 12-week Study of NFX-179 Gel in Subjects With Epidermal Nevi
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsored declined to proceed
Sponsor: Albert Chiou (Other)
Collaborators: NFlection Therapeutics, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Albert Chiou, Clinical Associate Professor, Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 60276
Record Dates: First submitted 2021-12-13; First posted 2022-01-19 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Epidermal Nevi; Nevus Sebaceus
MeSH Terms: conditions — Nevus, Sebaceous of Jadassohn

STUDY DESIGN:
Intervention Model Description: Open-label, all participants will apply NFX-179 gel for 12 weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Patients receiving NFX-179 Gel (Experimental): NFX-179 Gel 1.50% applied QD for 12 weeks
  Interventions: Drug: NFX-179 Gel 1.50%

INTERVENTIONS:
Drug: NFX-179 Gel 1.50% — Stanford University (Stanford) is studying a selective mitogen-activated protein kinase kinase (MEK) inhibitor (NFX-179) that has been chemically engineered for topical application to treat epidermal nevus syndromes (ENS).
  Preclinical studies evaluating topical application of NFX-179 to human nevus sebaceous explants demonstrated that NFX-179 can penetrate the tissue and suppress the p-ERK biomarker.
  It was also determined that NFX-179, when incubated with the tissues in medium, also suppressed ERK phosphorylation in human keratinocytic epidermal nevi. This clinical study is designed to evaluate the safety, tolerability, and clinical effect of NFX-179 Gel in Subjects with Epidermal Nevi.

SUMMARY:
This study of NFX-179 is an open-label study, evaluating safety, tolerability, pharmacodynamic activity, and the clinical effect in subjects with Epidermal Nevus(ENS). NFX-179 is formulated as a gel for topical administration. NFX-179 has been shown in animal studies and in human extracts to suppress p-ERK with systemic absorption of NFX-179 following topical application to be extremely low, based on serum values observed in animal studies.

Primary objectives:

* To determine the pharmacodynamic activity of NFX-179 Gel as defined by suppression of phospho-ERK (p-ERK) levels in Target EN in treatment group after 12 weeks of once-daily (QD) application
* To determine the safety and tolerability of treatment with NFX-179 Gel 1.50% applied QD for 12 weeks.

Secondary objectives:

-Clinical effect of NFX-179 Gel 1.5% defined as the percent change in EN volume after 12 weeks of QD application

DETAILED DESCRIPTION:
This is a 12-week clinical study to determine safety, tolerability, and clinical effect of NFX-179 Gel 1.50% Gel in subjects with EN.

At Visit 1 (Screening), the Investigator will select 1 Target EN lesion for treatment that meet the inclusion criteria. A biopsy tissue sample of the Target EN will be taken for histological confirmation of an EN diagnosis if required, to assess p-ERK levels and for genetic testing.

Subjects will be seen at Visit 2 for management of the Visit 1 biopsy wounds.

At Visit 3 (Baseline) eligible subjects will be provided study medication and start the 12-week, QD treatment period. Target EN assessments will be collected.

Subjects will be seen for treatment period visits, Visits 4-7, when Target EN assessments will be collected.

At Visit 8, subjects will be seen for the final treatment period visit. Target EN assessments, a biopsy sample for genetic testing and p-ERK levels will be. Subjects will start a 4-week no-treatment follow-up period.

Subjects will be seen at Visit 9, for management of the Visit 8 biopsy wound.

At Visit 10 (end of study), subjects will be seen for the final study visit and will be discharged from the study.

ELIGIBILITY:
Inclusion Criteria

In order to be eligible to participate in this study, all of the following criteria must be met:

1. Subject is at least 18 years of age
2. Subject must provide written informed consent prior to any study procedures
3. Subject has a Target Epidermal Nevi for treatment that:

   * Is a documented, biopsy proven, keratinocytic epidermal nevi (KEN) or nevus sebaceous (NS) or has a 3mm punch biopsy taken for histologic examination to determine KEN or NS status
   * Is a discrete lesion surrounded with at least 5mm of non-involved skin
   * Is not irritated
   * Does not have an active cutaneous infection
   * Has a Length ≥15mm
   * Has a surface area ≤100cm2
   * Has an Investigator's Lesion Assessment grade ≥2
   * Is located at an anatomical site that the subject can reach to apply the study medication
   * Has never been surgically treated
4. Subject is willing to have hair in the area surrounding the Target EN shaved, if necessary, to obtain photographs
5. Subject is willing to minimize exposure of the Target EN to natural or artificial ultraviolet radiation
6. Subject is willing to abstain from application of non-study topical prescription and over the counter medications to the Target EN during the study
7. Subject is willing to forego treatment of the Target EN, except protocol specified therapy, during the study
8. Female subjects who are women of childbearing potential must have a negative urine pregnancy test result and be willing to use a protocol approved, contraceptive method for the duration of the study.
9. Subject is willing and able to follow all study instructions and to attend all study visits.

No waivers to the inclusion criteria are permitted.

Exclusion Criteria A potential subject who meets any of the following criteria will be excluded from participation in this study:

1. Subject has applied any of the following topical products in the previous 30 days on or in proximity to the Target EN that, in the investigator's opinion, impairs evaluation of the Target EN or which exposes the subject to an unacceptable risk by study participation:

   * Topical glucocorticoid steroids
   * Topical retinoids (e.g., tazarotene, tretinoin, adapalene)
   * > 5% of an alpha-hydroxy acid (e.g., glycolic acid, lactic acid)
   * Fluorouracil
   * Imiquimod
2. The Target EN has ever been treated with a topical MEK inhibitor or a topical BRAF inhibitor
3. The Subject has used any of the following systemic medications in the noted time period:

   * Systemic retinoids (e.g., etretinate, isotretinoin) in the previous 90 days
   * Systemic MEK inhibitors in the previous 180 days
   * Systemic BRAF inhibitors in the previous 180 days
4. Subject has a history of hypersensitivity to any of the ingredients in the study medications
5. Subject has any know intercurrent illness or physical condition that would, in the investigator's opinion, impair evaluation of the Target EN or which exposes the subject to an unacceptable risk by study participation
6. Subject has, in the Investigator's opinion, a clinically relevant history of liver disease, including viral hepatitis, current alcohol abuse, or cirrhosis
7. Subject has a history of metastatic disease, or active cancer (excluding non-melanoma skin cancer, Stage I cervical cancer, ductal carcinoma in situ of the breast, or Stage 0 chronic lymphocytic lymphoma) within the previous 5 years
8. Subject has any condition (e.g., other skin conditions or diseases, metabolic dysfunction, physical examination findings, clinical laboratory findings) or situation (e.g., vacation, scheduled surgery) that would, in the Investigator's opinion, impair evaluation of the Target EN or which exposes the subject to an unacceptable risk by study participation
9. Subject has participated in an investigational drug trial in which administration of an investigational study medication occurred within the previous 30 days No waivers to the exclusion criteria are permitted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-06 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
The frequency of dermal safety and tolerability assessments including pain/burning, pruritus, erythema, edema, scabbing/crusting, and vesiculation/erosion | 12 weeks
  To determine the safety and tolerability of treatment with NFX-179 gel applied QD for 12 weeks of treatment.
The frequency of adverse events and serious adverse events as assessed by CTCAE v4.0 | 12 weeks
  To determine the safety and tolerability of treatment with NFX-179 gel applied QD for 12 weeks of treatment.

SECONDARY OUTCOMES:
Change in ILA (Investigator's Lesion Assessment) | 12 weeks
  Change in Investigator's Lesion Assessment after 12 weeks of QD application, assessed at screening, baseline, treatment period at week 2, 3, 4, and 8, and end of treatment at week 12.
Percent change in EN volume | 12 weeks
  Percent change in EN volume after 12 weeks of QD application as determined based on EN size derived from ruler measurements, and/or digital images from standardized photography performed at screening, baseline, treatment period at week 2, 3, 4, and 8, and end of treatment at week 12.

CONTACTS AND LOCATIONS:
Overall Officials: Albert S Chiou, MD, MBA, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Redwood City, California, United States

IPD SHARING:
Plan to Share IPD: No
We will only be sharing participant data with the sponsor, Nflection Therapeutics.